CLINICAL TRIAL: NCT04410497
Title: Silver Foam Dressing Superior to Porcine Xenograft in Pediatric Scalds: A Prospective Randomized Controlled Trial
Brief Title: Silver Foam Dressing Superior to Porcine Xenograft in Pediatric Scalds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Linkoeping (Other)
Responsible Party: Principal Investigator, Folke Sjoberg, Professor, University Hospital, Linkoeping
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DPS-2014
Record Dates: First submitted 2018-11-21; First posted 2020-06-01 (Actual); Last update posted 2020-06-01 (Actual); Status verified 2020-05

CONDITIONS: Burns Scald
Keywords: burns dressings healing

STUDY DESIGN:
Intervention Model Description: Prospective randomised trial were children, after Guardians written consent,are randomized to one of two dressings.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Porcine xenograft (Experimental): Conformité Européenne/European Conformity (CE)-marked dressing product used in clinical practise (Standard of care).
  Interventions: Other: Porcine xenograft (wound dressings)
- Silver foam (Active Comparator): Conformité Européenne/European Conformity (CE)- marked dressing product used in clinical practise
  Interventions: Other: Silver foam (wound dressings)

INTERVENTIONS:
Other: Porcine xenograft (wound dressings) — commercial porcine xenograft, derived from acellular dermis from porcine.
  Other Names: EZderm from Mölnlycke Healthcare AB, Gothenburg, Sweden
  Arms: Porcine xenograft
Other: Silver foam (wound dressings) — commercial silver containing foam dressing
  Other Names: Mepilex Ag from Mölnlycke Healthcare AB, Gothenburg, Sweden
  Arms: Silver foam

SUMMARY:
Prospective randomized trial where two dressings has been compared for partial thickness scald burns in children 6 months to 6 years.

DETAILED DESCRIPTION:
Aim: The aim of this study was to compare two different treatment regimes for children with partial-thickness scald burns. Burns were treated with either a porcine xenograft (EZderm®, Mölnlycke Health Care, Gothenburg, Sweden) or a silver foam dressing (Mepilex® Ag, Mölnlycke Health Care, Gothenburg, Sweden).

Methods: A prospective randomized clinical trial including 58 children admitted between May 2015 and May 2018 for partial-thickness scalds to The Burn Centre in Linkoping, Sweden. Primary outcome was time to wound closure. Secondary outcomes were pain, need of surgery, wound infection, length of hospital stay, required dressings changes, and labour time.

ELIGIBILITY:
Inclusion Criteria:

* Partial-thickness scald burns admitted within 72 hours of injury and with burns suitable for porcine xenograft according to the burn surgeon on duty were eligible and enrolled after (guardians) consenting to participate.

Exclusion Criteria:

* Children with other severe concomitant cutaneous trauma, skin disease, or children with a known hypersensitivity to silver.

Ages: 6 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 58 (Actual)
Dates: Start 2015-05-11 (Actual); Primary Completion 2018-05-08 (Actual); Study Completion 2018-05-08 (Actual)

PRIMARY OUTCOMES:
Time to complete wound closure | Evaluated 2-3 times per week until complete wound closure, approximatley 15-20 days after injury (injury-complete healing)
  Calculated from the date of injury to the date when the wound bed was assessed as completely reepithelialized with no necessity for further wound dressings other than a protective dressing against shearing, according to both the attending physician and nurse

SECONDARY OUTCOMES:
Pain (at wound site) | Evaluated before,during and after dressing changes, performed 2-3 times per week until complete wound closure, approximatley 15-20 days after injury.
  Pain is to evaluated by staff before, during and after wound dressing Changes using the Face, Legs, Activity, Cry, Consolability, behavioural pain scale (FLACC) is a five-category behavioral instrument where each category is scored on a scale of 0-2, resulting in a result between 0-10
Need of surgery | Evaluated at dressing changes, performed 2-3 times per week until complete wound closure, approximatley 15-20 days after injury.
  Evaluated as yes or no (surgery perfomered according to the medical record)
Burn wound infection | Evaluated at each dressing change; 2-3 times per week until complete wound closure, approximatley 15-20 days after injury.
  Children were diagnosed with burn wound infection by the burn surgeon and a consultant physician specialized in infectious diseases if fulfilling at least two of the following criteria based on American Burn Association definition of burn wound infection
  * Clinical signs such as localised pain and swelling, spreading erythema (redness), and heat at the affected site.
  * Surface wound swab culture presenting a minimum of 106 colony-forming units (CFU)/L (equivalent to the ABA definition of 105 CFU/g) [29].
  * Systemic signs of infection indicated as a rise of C-reactive protein (CRP) level (reference range < 10 mg/L for capillary sampling) together with increased body temperature exceeding 38 °C- 48 hours after injury where other sources of infection are excluded
Length of hospital stay | Evaluated after complete wound closure, approximatley 15-20 days after injury.
  number of days when the child received in hospital care (including readmissions)
number of dressing changes required | Evaluated at dressing changes, performed 2-3 times per week until complete wound closure, approximatley 15-20 days after injury.
  documented in CRF and in medical records
adverse events | Evaluated at dressing changes, performed 2-3 times per week until complete wound closure, approximatley 15-20 days after injury.
  any local reaction seen in or around wound during the time when study dressings were used
Minutes needed for application and removal of dressing | Evaluated at dressing changes, performed 2-3 times per week until complete wound closure, approximatley 15-20 days after injury.
  documented in CRF and in medical records

CONTACTS AND LOCATIONS:
Overall Officials: Johan Thorfinn, Ass.prof., Principal Investigator — Linkoping Burn Centre, University hospital of Linkoping, Sweden
Locations (1):
- The Burn Centre at Linköping University Hospital,, Linköping, Sweden

IPD SHARING:
Plan to Share IPD: No
only if asked for